CLINICAL TRIAL: NCT04536740
Title: Effect of Pulsed Dye Laser on Photodynamic Therapy of Port-Wine Stains: a Single Center, Perspective, Paralled, Controlled Clinical Trial
Brief Title: Effect of Pulsed Dye Laser on Photodynamic Therapy of Port-Wine Stains
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gang Ma (Other)
Responsible Party: Sponsor-Investigator, Gang Ma, Associate Professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Organization: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SH9H-2020-T290-1
Record Dates: First submitted 2020-08-22; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Port-Wine Stain
Keywords: pulsed dye laser; photodynamic therapy
MeSH Terms: conditions — Port-Wine Stain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PDL-treated PWS (Other): PWS treated with PDL before will be treated with PDT
  Interventions: Device: PDT treatment device
- without treatment PWS (Experimental): PWS without treatment before will be treated with PDT
  Interventions: Device: PDT treatment device

INTERVENTIONS:
Device: PDT treatment device — All patients will be treated under general anesthesia. After carefully covering the normal skin, hematoporphyrin monomethyl ether (HMME; Shanghai Fudan-Zhangjiang Bio-Pharmaceutical, Shanghai, China) was i.v. transfused at a dose of 5 mg/kg for 20 min at a constant rate. Five to 10 min after the onset of HMME transfusion, continuous irradiation at 532 nm (532-nm light-emitting diode green-light therapeutic apparatus; Wuhan Yage Optic and Electronic Technique, Wuhan, China) was applied with a power density of 80- 95 mW/cm2 for 20-30 min. Concomitant forced air cooling was applied during irradiation for epidermal protection. Post-treatment skin cooling was performed by intermittent application of ice packs over a 3-day period, to minimize pain and potential thermal damage. To prevent the effects of photosensitivity, patients were instructed to avoid exposure to strong light for at least 14 days after treatment.
  Other Names: light-emitting diode green-light therapeutic apparatus

SUMMARY:
Port-wine stain (PWS) is a congenital capillary malformation with an incidence of 3-5/1000 newborns and grows commensurately with the affected individual.

Although PDL treatment can significantly lighten and reduce most PWS lesions, 20% of cases show little improvement after treatment. Our previous researches suggested that PDT may be a beneficial option for PWS cases that are resistant to multiple PDL treatments.

In this study, a single center, prospective, parallelled, controlled study was conducted to compare the efficacy of PDT on PWS treated with standard PDL and those without any treatment.

DETAILED DESCRIPTION:
Port-wine stain (PWS) is a congenital capillary malformation characterized by ectatic capillaries and postcapillary venules located predominantly in the papillary and mid-reticular layers of the dermis. It has an incidence of 3-5/1000 newborns and grows commensurately with the affected individual.

Pulsed dye laser (PDL) of 585 and 595 nm is considered to be the gold standard for treating PWS. Although PDL treatment can significantly lighten and reduce most PWS lesions, 20% of cases show little improvement after treatment. This ratio therefore represents a relatively large number of patients who may benefit from an alternative treatment modality.

Vascular-targeted photodynamic therapy (PDT) has been used to treat PWS since the 1990s. In 1990, Orenstein et al. used a chicken comb model to show that PDT can treat hypervascular dermal lesions while leaving the normal overlying epidermis completely intact. The use of vascular-targeted PDT for treating PWS was first described in 1991. PDT can theoretically target ectatic capillaries of all diameters and, in contrast to PDL, can induce vascular damage deeper in the dermis, with a considerably reduced risk of epidermal necrosis due to its vascular-selective characteristics. Previous studies have also demonstrated that PDT is an effective and safe means of improving the appearance of PWS.

Our previous researches suggested that PDT may be a beneficial option for PWS cases that are resistant to multiple PDL treatments.Therefore, the choice of early treatment for PWS is very important . The effect of PDL therapy on the follow-up photodynamic treatment of PWS unknown.

In this study, a single center, prospective, parallelled, controlled study was conducted to compare the efficacy of PDT on PWS treated with standard PDL and those without any treatment. Our objectis to explore whether the previous PDL treatment will affect the efficacy of the follow-up PDT on PWS, so as to provide early treatment options for children with PWS.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1-14 years who met the criteria for diagnosis of port-wine stain in The International Society for the Study of Vascular Anomalies（ISSVA);
* Patients in the untreated group had never received any treatment;
* Patients in the PDL-treated group received at least five 595 nm pulse dye laser (PDL) treatment (Vbeam laser; candela Corp., Boston, MA), The time interval between
* Photodynamic therapy and the last pulse dye laser treatment was at least 3 months;
* There were complete medical records, standard photos and test records before and after treatment;
* After fully understanding the treatment plan and risks, patients voluntarily signed the informed consent and was willing to accept clinical trials and cooperate with follow-up.

Exclusion Criteria:

* Original infection, eczema, ulcers in the lesion site; The patient has a history of seizures in the last six months or the condition is not under control;
* Hypersensitivity to porphyrins, hypersensitivity constitution;
* Scar constitution;
* A history of heavily UV exposure in the last 3 months;
* With abnormal electrocardiogram, heart disease, liver damage, pregnancy or other underlying diseases that may affect treatment;
* Patients are participating in other clinical trials.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Visual evaluation | Change from Baseline Visual evaluation at 3 months after PDT treatment
  Standard digital photographs were obtained using consistent camera settings (EOS 80D; Canon, Tokyo, Japan), light conditions and patient positions. Three independent, blinded assessors qualitatively assessed color blanching

SECONDARY OUTCOMES:
Chromameter evaluation | Change from Baseline Chromameter evaluation at 3 months after PDT treatment
  Blanching of the PWS lesions was evaluated using a SkinColorCatch" chromameter (Delfin Technologies, Kuopio, Finland).

IPD SHARING:
Plan to Share IPD: Undecided